CLINICAL TRIAL: NCT01983124
Title: A Phase II Single-arm Study for the Treatment After Recurrence of Advanced Melanoma Patients Harboring the V600BRAF Mutation and Pretreated With Vemurafenib, With the Association of Vemurafenib Plus Fotemustine.
Brief Title: Vemurafenib + Fotemustine to Treat Advanced Melanoma Patients With V600BRAF Mutation Recurred While on Vemurafenib
Acronym: BeyPro1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Paola Queirolo (Other)
Collaborators: Istituto Nazionale per lo Studio e la Cura dei Tumori (Other)
Responsible Party: Sponsor-Investigator, Paola Queirolo, MD, IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Organization: IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-004172-18
Record Dates: First submitted 2013-11-06; First posted 2013-11-13 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Malignant Melanoma Stage IV
Keywords: Advanced Melanoma
MeSH Terms: conditions — Melanoma | interventions — fotemustine; Vemurafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fotemustine + Vemurafenib (Experimental): Fotemustine 100 mg/m2 q21 + Vemurafenib gelatin capsules supplied as 240-mg strengths. Vemurafenib will be administered continuous oral dosing at 960 mg twice daily or dose administered at time of disease progression with Vemurafenib previous treatment.
  Interventions: Drug: Fotemustine + Vemurafenib

INTERVENTIONS:
Drug: Fotemustine + Vemurafenib — Fotemustine 100mg/m2 IV on day 1 of each 21 day cycle. Number of cycles: until progression or unacceptable toxicity.
  Vemurafenib administered continuous oral dosing 960 mg twice daily or dose administered at time of progression since progression or unacceptable toxicity.
  Other Names: Fotemustine; Zelboraf

SUMMARY:
The purpose of this study is to evaluate the activity of Vemurafenib in combination with Fotemustine in Patients with unresectable Stage IV melanoma harboring V600 BRAF mutation who recurred while in treatment with Vemurafenib. In addition the feasibility and safety profile of prolonging treatment of this drugs combination will be assessed.

DETAILED DESCRIPTION:
Patients are treated with Fotemustine 100 mg/m2 q21 + Vemurafenib. Vemurafenib will be administered continuous oral dosing at 960 mg twice daily or dose administered at time of disease progression with Vemurafenib previous treatment (720 or 480 mg).Treatment will be continued until progression or unacceptable toxicity. The Progression-free survival will be assessed as primary endpoint, other outcomes(i.e., incidence of grade III-IV toxicity, Disease Control Rate, and Overall Survival) will be considered secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed melanoma harboring the V600 mutation
* Unresectable Stage IV melanoma
* At least 18 y of age
* Eastern Cooperative Oncology Group (ECOG) performance status of <2
* In progression during treatment with Vemurafenib
* At least 2 weeks since the last radiotherapy treatment
* Life expectancy >12 weeks
* Clinical laboratory values at screening defined as follow: lactate dehydrogenase (LDH) < 2.0 x upper limit of normal (ULN), Hemoglobin >9 g/dL, Absolute neutrophil count 1500/mm3, Platelet count >100,000/mm3, Creatinine <1.5 mg/dL (NOTE: If creatinine is >1.5 mg/dL, subject is eligible if creatinine clearance > 60 mL/min using the Cockgroft-Gault equation), Total bilirubin <1.5 x ULN, Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) <2.5 x ULN
* Negative serum pregnancy test within 7 days prior to commencement of dosing in premenopausal women. Women of non-childbearing potential may be included if they are either surgically sterile or have been postmenopausal for ≥ 1 year
* Fertile men and women must use an effective method of contraception
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Female subjects who are pregnant or nursing
* Female subjects of childbearing potential or males not using or not willing to use two forms of effective contraception
* Any of the following within the 6 months prior to randomization: myocardial infarction, severe/unstable angina, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, pulmonary embolism, hypertension not adequately controlled by current medications
* Concurrent administration of any anti-cancer therapies (e.g. chemotherapy, other targeted therapy, experimental drug, etc) other than those administered in this study
* Known hypersensitivity to Vemurafenib or another BRAF inhibitor
* History of congenital long QT syndrome, history or presence of clinically significant ventricular or atrial dysrhythmias ≥ Grade 2 (NCI Common Toxicity Criteria for Adverse Effects (CTCAE) Version 4.0
* Corrected QT (QTc) interval ≥ 500 msec at baseline
* Uncontrolled medical illness (such as infection requiring treatment with intravenous (IV) antibiotics)
* Has had surgery within 2 weeks (1 week for minor surgery, eg, procedures requiring only local anesthetics) prior to the first dose of study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-02; Primary Completion 2014-04 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 6 months
  To assess activity of vemurafenib in combination with fotemustine, in patients harboring the V600BRAF mutation and recurred while on treatment with Vemurafenib.

SECONDARY OUTCOMES:
Incidence of Grade 3-4 toxicities (any type) | 6 months
Rate, duration of response and proportion of patients with duration of response lasting > 24 weeks | 6 months
Disease control rate; | 6 months
Time to progression of brain metastases (BM), Including incidence of BM in pts free from BM at the time of enrolment | 6 months
Overall survival (OS). | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Paola Queirolo, MD, Principal Investigator — IRCCS AOU San Martino IST
Locations (2):
- Italy (2):
  - Paola Queirolo, Genova
  - Istituto Nazionale per lo Studio e la Cura dei Tumori "G.Pascale", Napoli

REFERENCES:
- [Derived] Queirolo P, Spagnolo F, Picasso V, Spano L, Tanda E, Fontana V, Giorello L, Merlo DF, Simeone E, Grimaldi AM, Curvietto M, Del Vecchio M, Bruzzi P, Ascierto PA. Combined vemurafenib and fotemustine in patients with BRAF V600 melanoma progressing on vemurafenib. Oncotarget. 2016 Jul 13;9(15):12408-12417. doi: 10.18632/oncotarget.10589. eCollection 2018 Feb 23. PMID 29552321